CLINICAL TRIAL: NCT00843596
Title: Surgical Bleeding Control of Extra-corporeal Circulation (ECC) by Vacuum Devices
Acronym: HEMOCARD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AdministrateurCIC (Other)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 0809
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Bleeding
Keywords: cardiac surgery requiring ECC
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vacuum device - suction cup (Experimental)
  Interventions: Procedure: cardiac surgery requiring ECC

INTERVENTIONS:
Procedure: cardiac surgery requiring ECC — the vacuum device is left on the 2 wounds (caused by the ECC cannulas) for 15 min (possible a second time of 15 min : 30 min max.)

SUMMARY:
the purpose of this study is to show that the vacuum control surgical bleeding helps stop bleeding extraMD (MD: Medical Device) at the orifice of the retrograde cannulation during a heart with Extra-corporeal circulation (ECC),

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old
* patient affiliated to social security or similarly regime
* patient sent to hospital for cardiac surgery requiring ECC

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Person participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Persistence or absence of bleeding extraMD at the orifice of the retrograde cannulation when the suction cup is in place. | 20-30 min

SECONDARY OUTCOMES:
Persistence or absence of bleeding intraMD at the orifice of the retrograde cannulation when the suction cup is in place. | 20-30 min
Persistence or absence of bleeding at the orifice of the retrograde cannulation when the vacuum was removed. | 20-30 min
Persistence or absence of bleeding extraMD at the orifice of the aortic purge when the suction cup is in place. | 20- 30 min
Persistence or absence of bleeding extraMD at the orifice of the aortic purge when the suction cup is in place. | 20 -30 min
Persistence or absence of bleeding at the orifice of the aortic purge when the vacuum was removed. | 20 -30 min

CONTACTS AND LOCATIONS:
Overall Officials: Dominique BLIN, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- UniversityHospitalGrenoble, Grenoble, France